CLINICAL TRIAL: NCT00267267
Title: Phase 3, Open-Label, Multi-Center, Double-Blind, Randomized, Parallel Group Study Efficacy and Safety of Fixed Combination Torcetrapib/Atorvastatin, Administered Once Daily (QD) Compared to Fixed Combination Ezetimibe/Simvastatin for 6 Weeks in Subjects With Dyslipidemia.
Brief Title: A Clinical Trial Comparing Torcetrapib/Atorvastatin to Ezetimibe/Simvastatin In Subjects With A Cholesterol Disorder.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091035
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2006-12

CONDITIONS: Hyperlipidemia; Dyslipidemia
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias | interventions — torcetrapib; Atorvastatin; Ezetimibe, Simvastatin Drug Combination

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: ezetimibe/simvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

Cholesterol levels will be measured over six weeks in subjects being treated with two different kinds of combination cholesterol medications to see how the different treatments compare to one another.

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Specific LDL-C levels based on CHD risk after a six-week washout period.

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors.
* Subjects requiring systemic steroids
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1784
Dates: Start 2006-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C and HDL-C from baseline, after six weeks of treatment.

SECONDARY OUTCOMES:
Changes in other lipid parameters and other biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (103):
- United States (103):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Los Altos, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Rose, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Westlake Village, California
  - Pfizer Investigational Site, Golden, Colorado
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Atlantis, Florida
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Daytona Beach, Florida
  - Pfizer Investigational Site, DeFuniak Springs, Florida
  - Pfizer Investigational Site, Destin, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Aurora, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Newton, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Edgewood, Kentucky
  - Pfizer Investigational Site, Erlanger, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Ayer, Massachusetts
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Bloomfield Hills, Michigan
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Brooklyn Center, Minnesota
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, Manchester, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Cooperstown, New York
  - Pfizer Investigational Site, Endwell, New York
  - Pfizer Investigational Site, Lewiston, New York
  - Pfizer Investigational Site, Manlius, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Monroe, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Wilmington, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Fairview Park, Ohio
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Doylestown, Pennsylvania
  - Pfizer Investigational Site, Harleysville, Pennsylvania
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Sayre, Pennsylvania
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Simpsonville, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Selmer, Tennessee
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Bountiful, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Newport News, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Spokane, Washington